CLINICAL TRIAL: NCT01302561
Title: Protocol 2: Galactooligosaccharide, Immune Strength, and Digestive Health in Older Adults Over Cold and Flu Season
Brief Title: Galactooligosaccharide, Immune Strength, and Digestive Health in Older Adults Over Cold and Flu Season
Acronym: GOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GTC Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 355-2010
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: adults; fiber; cold; flu; immune function; microbiota
MeSH Terms: conditions — Common Cold; Influenza, Human | interventions — Sucrose; 4'-galactooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator)
  Interventions: Dietary Supplement: Sucrose
- Galactooligosaccharide 5 g (Experimental)
  Interventions: Dietary Supplement: Galactooligosaccharide

INTERVENTIONS:
Dietary Supplement: Sucrose — 5 g of sucrose twice daily for 24 weeks
  Arms: Sugar Pill
Dietary Supplement: Galactooligosaccharide — 2.5 g galactooligosaccharide plus 2.5 g sucrose twice daily for 24 weeks
  Arms: Galactooligosaccharide 5 g

SUMMARY:
The purpose of this research study is to determine whether a functional fiber, galactooligosaccharide, can help maintain immune strength and digestive health in free-living older adults. It is hypothesized that older adults consuming the fiber daily for 24 weeks over cold and flu season will have more healthy days due to a proliferation of beneficial bacteria within the colon which alters cytokine production and enhances natural killer cell function. Immune and gastrointestinal health will be evaluated via daily questionnaires obtained from 80 participants and from the collection of blood and fecal samples.

DETAILED DESCRIPTION:
A prospective, randomized, parallel, double-blind, placebo controlled trial will be used. Healthy older adults will be recruited from the Gainesville area via direct mailing, flyers, list servs, presentations to clubs/organizations/church groups, social networks, etc. Informed consent will be obtained and once the informed consent is signed the inclusion/exclusion form will be reviewed to determine whether a subject qualifies for the study.

Prior to randomization, height, weight, age, and a stool sample will be obtained. On the day of randomization, blood will be drawn and saliva will be collected for baseline immune function studies from all subjects who qualify based on the final criteria (i.e., cannot have a cold on the day of randomization).

Subjects will be stratified based on body mass index and age and randomized via sealed envelope to the treatment (5 g GOS) or placebo groups (n=40/group). The fiber will be provided in small packets containing 2.5 g of fiber and 2.5 g sucrose (treatment) or 5 g of sucrose (placebo). Subjects will be instructed to add the contents of the packet to coffee, tea, water, milk, or other non-carbonated drink, hot cereal or pudding and mix well. Subjects will be told to consume two packets per day and maintain a daily study log. The daily questionnaire will ask about intake of the fiber, cold symptoms, and general health (i.e., new medications, doctor visits).

Between weeks two and three of the intervention, a second stool sample will be obtained. After three weeks of the intervention, subjects will receive the influenza vaccination and blood and saliva will be collected for immune function studies. Two weeks postvaccination (i.e., 5 weeks of intervention), blood and saliva will be collected for immune function studies. Subjects will continue the intervention and maintain daily logs for a total of 24 weeks. Subjects will also be asked to complete a questionnaire on a monthly basis regarding gastrointestinal symptoms and typical level of exercise.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* willing to complete daily and monthly questionnaires
* willing to receive the fall influenza vaccination as part of the study protocol
* willing to provide 3 blood samples, 3 saliva samples, and 2 stool samples and answer a food frequency questionnaire over the course of the study
* willing to discontinue any immune-enhancing dietary supplements ( e.g., prebiotics and fiber supplements, probiotics, echinacea, fish oil, vitamin E >100% of the RDA or >15 mg/day)
* willing to take the study fiber for 24 weeks
* willing to provide a social security number to receive study payment Note: the subject can still participate if unwilling to provide SS#, but no financial reimbursement can be provided.
* had a cold in the last 12 months
* able to take foods and the study fiber without the aid of another person.
* eligible and willing to receive the influenza vaccine for the current year. That is, you cannot have already received an influenza vaccine for the 2010/2011 season prior to receiving it from the study

Exclusion Criteria:

* current smoker
* chronic allergies involving the upper respiratory tract (Chronic = taking allergy medicine daily)
* taking any medication for constipation or diarrhea
* currently taking any anti-inflammatory drugs on a regular basis
* currently treated for Alzheimer's disease
* allergy to milk or a serious allergy to eggs (note lactose intolerance should not be a problem because 1 fiber packet contains only 0.3 g of lactose whereas 1 cup of milk contains 12.8 g of lactose)
* currently being treated for any known illnesses or conditions that may impact perceived health such as HIV/AIDS, immune modulating diseases (autoimmune, hepatitis, cancer, etc.), diabetes, kidney disease, gastrointestinal diseases (gastric ulcers, Crohn's, ulcerative colitis, etc.)
* received chemotherapy or other immune suppressing therapy within the last year
* received antibiotic therapy in the past two months
* receiving supplemental oxygen

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Percentage of days without cold/flu symptoms | Measured Daily for 24 weeks
  * Average number of cold symptoms [Nasal Symptoms (Running Nose, Stuffed nose, Blowing the Nose, Yellow Secretion, Bloody Secretion), Pharyngeal Symptoms (Scratchy Throat, Sore Throat, Hoarseness), Bronchial Symptoms (Cough, Secretion, Yellow Secretion), Headache, Achiness (Muscle Pain), Conjunctivitis (Reddish Eyes), Fatigue, Ear Discomfort and Stiffness/Chills]
  * Average sum of symptom intensity
  * Cold symptom score (sum of symptom intensity scores)

SECONDARY OUTCOMES:
Digestive Health | Measured Monthly for 24 weeks
  * Symptoms (gas, bloating, diarrhea, etc.)
  * Bowel habits (bowel movement frequency and consistency)
Immune Function | Measured at baseline, week 3 and week 5 of the intervention
  * Leukocyte phenotype and function
  * Peripheral blood mononuclear cell cytokine production to mitogens
  * Serum acute phase proteins, cytokines, endotoxin, and immunoglobulin
  * Salivary and fecal sIgA
Microbiota Study | Measured at baseline and between weeks 2 and weeks 3 of intervention
  * Microbial diversity measured by DGGE profiling (detect large distortions)
  * qPCR to quantify changes in Lactic Acid Bacteria and Bifidobacteria (beneficial changes)
  * 16S rRNA sequencing (454) to identify treatment effects on specific bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States